CLINICAL TRIAL: NCT02959242
Title: Dresden Glaucoma and Treatment Study: Analysis to Assure the Quality of Follow-up and Therapy of Glaucoma Patients in a Tertiary University Hospital Glaucoma Service.
Brief Title: Dresden Glaucoma and Treatment Study (DGTS)
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. Karin Pillunat, Dr. med., Technische Universität Dresden
Other Study IDs: DGTS
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Glaucoma; Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Glaucoma, Low Tension
Keywords: Follow-up intervals; Treatment Efficiency; Laser Therapy; Glaucoma Surgery; Minimal Invasive Glaucoma Surgery (MIGS)
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assure the quality of follow-up and treatment, data of glaucoma patients are stored and evaluated after anonymisation.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the quality of follow-up and treatment by means of consecutive data collection and anonymised analysis of all glaucoma patients of a tertiary university hospital glaucoma service.

Parameters being analyzed are:

Age, sex, refraction, family history, known duration of glaucoma, highest intraocular pressure before treatment, systemic and topical medication, previous ocular surgery.

24h Goldmann-applanation tonometry, biomicroscopy, gonioscopy, Heidelberg Retinal Tomograph (HRT), glaucoma diagnosis with Scanning-Laser-Polarimetry (GDx), optical coherence tomography (OCT), Pentacam, Ocular Response Analyzer (ORA), Corvis ST (Corneal Visualization with the Scheimpflug Technology), perimetry

ELIGIBILITY:
Inclusion Criteria:

* manifest glaucoma, ocular Hypertension, glaucoma suspect

Exclusion Criteria:

* under 18 years of age, corneal diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Glaucoma patients attending a tertiary University Hospital glaucoma Service.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2006-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Follow-up intervals | 20 years
  To find the best follow-up intervals for glaucoma patients.

SECONDARY OUTCOMES:
Assessment of treatment quality | 20 years
  What is the best treatment option for the individual patient?
Assessment of intraocular pressure-lowering efficacy and number of participants with treatment-related adverse events as assessed by CTCAE v4.0 of glaucoma laser therapy | 20 years
  Diurnal intraocular pressure, best corrected visual acuity, visual fields
Assessment of intraocular pressure-lowering efficacy and number of participants with treatment-related adverse events as assessed by CTCAE v4.0 of glaucoma laser therapy of glaucoma surgery | 20 years
  Diurnal intraocular pressure, best corrected visual acuity, visual fields

CONTACTS AND LOCATIONS:
Overall Officials: Lutz E Pillunat, MD, PhD, Study Director — Medical faculty of the Technical University of Dresden, Germany
Locations (1):
- University Eye Hospital, Medical Faculty, Technical University Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data are only shared between researchers of our Institute.

REFERENCES:
- [Derived] Pillunat KR, Herber R, Jamke M, Jasper CS, Haase MA, Manseck AS, Pillunat LE. Early Results of Preserflo MicroShunt for Primary Open Angle Glaucoma in White Patients. J Glaucoma. 2025 Feb 1;34(2):103-113. doi: 10.1097/IJG.0000000000002509. Epub 2024 Oct 11. PMID 39401481
- [Derived] Jamke M, Herber R, Haase MA, Jasper CS, Pillunat LE, Pillunat KR. PRESERFLO MicroShunt versus trabeculectomy: 1-year results on efficacy and safety. Graefes Arch Clin Exp Ophthalmol. 2023 Oct;261(10):2901-2915. doi: 10.1007/s00417-023-06075-4. Epub 2023 May 3. PMID 37133501
- [Derived] Pillunat KR, Kocket GA, Herber R, Jasper CS, Lenk J, Pillunat LE. Efficacy of selective laser trabeculoplasty on lowering intraocular pressure fluctuations and nocturnal peak intraocular pressure in treated primary open-angle glaucoma patients. Graefes Arch Clin Exp Ophthalmol. 2023 Jul;261(7):1979-1985. doi: 10.1007/s00417-022-05897-y. Epub 2022 Nov 23. PMID 36418515